CLINICAL TRIAL: NCT04465994
Title: Comparison of Mid-term Curative Effect After Primary Repair Versus Gastrocnemius Turn-down Flaps of Acute Achilles Tendon Rupture
Brief Title: Comparison of Primary Repair Versus Gastrocnemius Turn-down Flaps of Acute Achilles Tendon Rupture
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019465
Record Dates: First submitted 2020-06-27; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Acute Rupture of Achilles Tendon (Disorder)
Keywords: Achilles Tendon; Acute injury; Primary repair; gastrocnemius turn-down flaps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- primary repair: Patients with acute achilles tendon ruptures who received the treatment of primary repair.
- gastrocnemius turn-down flaps: Patients with acute achilles tendon ruptures who received the treatment of gastrocnemius turn-down flaps.
  Interventions: Procedure: gastrocnemius turn-down flaps

INTERVENTIONS:
Procedure: gastrocnemius turn-down flaps — We classified the patients with acute achilles tendon rupture by type of surgery. The group who received the gastrocnemius turn-down flaps is the intervention group.
  Groups: gastrocnemius turn-down flaps

SUMMARY:
This retrospective study includes 74 patients with acute Achilles tendon rupture from March 2012 to September 2018, aiming to compare the mid-term curative effect of primary repair and gastrocnemius turn-down flaps and guide clinical decision.

DETAILED DESCRIPTION:
Objective: To explore the surgical methods and observe the med-term curative effect of primary repair and gastrocnemius turn-down flaps for acute Achilles tendon rupture, so as to guide clinical decision. Methods: This retrospective study includes 74 patients with acute Achilles tendon rupture from March 2012 to September 2018, whose surgeries was completed by the sponsor with either primary repair or gastrocnemius turn-down flaps. The recovery and motor function of the patients were followed up by outpatient clinic and telephone at 3 months, 6 months, 12 months and 24 months after operation, respectively, so as to statistically analyze the med-term curative effects of two surgeries. Specific indicators include: Visual Analogue Scale, American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score, The Victorian Institute of Sport Assessment-Achilles, The Achilles tendon Total Rupture Score, the Tegner Activity Score, Biodex isokinetic dynamometer system, Postoperative rehabilitation index and complications.

ELIGIBILITY:
Inclusion Criteria:

* history of Achilles tendon injury
* within two weeks of injury
* inability to single heel rise
* more than one year of follow-up
* age under 65

Exclusion Criteria:

* open Achilles tendon rupture
* Achilles tendon terminal disease
* rerupture of Achilles tendon
* history of local corticosteroid injection around the Achilles tendon
* accompanied by fracture, vascular or nerve damage
* not available for regular follow-up

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study includes 74 patients with acute Achilles tendon rupture from March 2012 to September 2018, including 68 male patients and 6 female patients. The average age is 36 years.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
change of Visual Analogue Scale | from pre-surgery to two years after surgery
  The Visual Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. The minimum and maximum values of VAS are 10 and 0, respectively. And higher scores mean a worse outcome.
change of American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score | from pre-surgery to two years after surgery
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). The minimum and maximum values of AOFAS are 100 and 0, respectively. And higher scores mean a better outcome.
change of The Victorian Institute of Sport Assessment-Achilles | from pre-surgery to two years after surgery
  The VISA-A questionnaire displayed construct validity when used in two populations of patients with Achilles tendinopathy and control subjects. The questionnaire avoids the redundant components of non-specific scoring systems such as that developed for hind foot problems by the American Orthopaedic Society, and those devised for Achilles tendon rupture. Results range from 0 to 100, where 100 represents the perfect score.
change of The Achilles tendon Total Rupture Score | from pre-surgery to two years after surgery
  The VISA-A questionnaire displayed construct validity when used in two populations of patients with Achilles tendinopathy and control subjects. The questionnaire avoids the redundant components of non-specific scoring systems such as that developed for hind foot problems by the American Orthopaedic Society, and those devised for Achilles tendon rupture. Results range from 0 to 100, where 100 represents the perfect score.
change of the Tegner Activity Score | from pre-surgery to two years after surgery
  The Tegner activity scale was first described in 1985 and initially designed for physician administration after ACL and meniscal injuries. To date, the Tegner activity score has been a frequently used patient-administered activity rating system for patients with various knee disorders. The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Biodex | through study completion, an average of 2 years
  Biodex isokinetic dynamometer system

SECONDARY OUTCOMES:
complications | through study completion, an average of 2 years
  rerupture, infection, wound scar

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No